CLINICAL TRIAL: NCT03155100
Title: Phase 2 Study of Carfilzomib + Elotuzumab + Dexamethasone for Relapsed or Progressed Multiple Myeloma After 1-3 Prior Treatment Lines
Brief Title: Carfilzomib + Elotuzumab + Dexamethasone for Relapsed Multiple Myeloma After 1-3 Prior Treatment Lines
Acronym: KEd
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raija Silvennoinen (Other)
Collaborators: Amgen (Industry); Bristol-Myers Squibb (Industry); Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Sponsor-Investigator, Raija Silvennoinen, Principal Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMSG#24/15; 2016-001178-13 (EudraCT Number)
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma in Relapse
MeSH Terms: interventions — carfilzomib; Proteasome Inhibitors; elotuzumab; Antibodies, Monoclonal; Dexamethasone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carfilzomib, elotuzumab, dexamethasone (Experimental): Carfilzomib 70 milligram(mg)/m2 iv (56 mg/m2 for first five patients for cycles 1-2) once weekly, on days 1, 8 and 15 (cycles 1-8), from cycle 9 on days 1 and 15 until progression or toxicity; elotuzumab 10 mg/kg iv on days 1,8,15 for cycles 1-2, on days 1and 15 from cycle 3 until progression or toxicity; dexamethasone 40 mg weekly (shared to po and iv)
  Interventions: Drug: Carfilzomib for Inj 60 milligram (MG); Drug: Elotuzumab 400 MG; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib for Inj 60 milligram (MG) — All patients will have similar effective study drug combination; karfilzomib plus elotuzumab plus dexamethasone
  Other Names: Proteasome inhibitor
Drug: Elotuzumab 400 MG — All patients will have similar effective study drug combination; karfilzomib plus elotuzumab plus dexamethasone
  Other Names: Monoclonal antibody
Drug: Dexamethasone — All patients will have similar effective study drug combination; karfilzomib plus elotuzumab plus dexamethasone
  Other Names: Steroid

SUMMARY:
The main aim of this study is to assess the ORR with a new drug combination, carfilzomib (CAR) + elotuzumab (ELO) + dexamethasone (CAR-ELO-Dex).

DETAILED DESCRIPTION:
This Nordic Myeloma Study Group study is a phase 2 study for advanced multiple myeloma (MM) patients below 75 years of age. The main aim of this study is to assess the overall response rate (ORR) with a new drug combination, carfilzomib + elotuzumab + dexamethasone (CAR-ELO-Dex). Even if this is not a randomized study rough comparisons can be done with earlier reports of different regimens in the same clinical situation. In addition, safety assessment is of critical importance for a new regimen. A modern concept is to study the depth of complete responses (CR) with a sensitive multiparameter flow cytometry (MFC) method for minimal residual disease (MRD) assessment - an endpoint that is mostly lacking in previous studies for this patient population. We assume that treatment with this new combination of CAR + ELO + Dex will produce at least as good responses as the most efficient regimens so far used in this clinical situation, and there will be a substantial proportion of CR responses with MRD-negativity which can be regarded as an indicator of high-level treatment efficacy and which gives a good basis for comparisons of treatment efficacy between different study regimens in future.

The target population of the study is the patients who have relapsed or progressed after 1 to 3 prior treatment lines in which PI (bortezomib and/or ixazomib) and/or lenalidomide have been included. The primary endpoint is overall response rate while the secondary endpoints include complete remission, duration of response, assessment of the depth (quality) of CR with MRD measurement by flow cytometry, estimation of progression free survival (PFS) and time to next treatment, and evaluation of adverse events and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at the age of 18 to below 75 years with the life expectancy of at least three months.
2. Prior confirmed diagnosis of multiple myeloma and measurable disease in blood or urine with at least one of the following: Serum M-protein ≥ 5g/l, Urine M-protein ≥ 200 mg/24 hours, In subjects without detectable serum or urine M-component, serum free light chain (S-FLC) > 100 ml/l (involved light chain) and an abnormal serum kappa/lambda ratio
3. Relapse or progression after 1 to 3 prior treatment lines, which have included proteasome inhibitors (bortezomib, carfilzomib and/or ixazomib) and/or lenalidomide. Refractoriness to bortezomib, ixazomib and/or lenalidomide is allowed in the preceding cycle. Patients with previous autologous transplantation can be included.
4. Need of treatment of relapse or progression: IMWG criteria for relapse/progression (paraprotein or hypercalcemia, renal insufficiency, anemia, bone disease (CRAB) criteria or both). (Appendix 5)
5. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.
6. Females of childbearing potential (FCBP) must have a confirmed negative serum pregnancy test within the 7 days prior to inclusion
7. Females of childbearing potential must use one effective method of contraception and their partners condom during the study and for 120 days following the last study drug treatment dose and male subjects who are sexually active with FCBP must agree to use condom during the study and for 180 days following the last study drug treatment dose.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2, or Karnofsky at least 60.
9. Patients must meet the following adequate organ and bone marrow function within 21 days prior to inclusion:

   * Absolute neutrophil count (ANC) 1,000/mm3 (≥ 1.0 x 109/L) and platelet count 75 x 109/L. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment. Granulocyte growth factors are allowed to meet the inclusion criteria.
   * Hemoglobin (Hb) ≥ 80 g/l (use of erythropoietin and red blood cell transfusions allowed by institutional guidelines, however the most recent red blood cells (RBC) may not have given within 7 days prior to obtaining screening Hb
   * Total bilirubin < 1.5 times the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 times the ULN.
   * Calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault estimation of creatinine clearance (CRcl): CRcl (mL/min) = (140 - age) x (weight [kg]) / 72 x (serum creatinine [mg/dL]); for females, multiply by 0.85 (Cockcroft 1976, Luke 1990)
10. Patient must be willing and able to adhere to the study protocol visit schedule and other protocol requirements.
11. Negative pregnancy test at inclusion if applicable

Exclusion criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Major surgery within 28 days before enrollment.
3. Radiotherapy within 14 days before enrollment, but if the involved field is small, 7 days will be considered a sufficient interval before onset of the treatment.
4. Glucocorticoid therapy within the 14 days prior to inclusion that exceeds a cumulative dose of 160 mg dexamethasone or 1000 mg prednisone.
5. Central nervous system involvement.
6. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
7. Active congestive heart failure (NYHA III-IV) (Appendix 3), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, acute diffuse infiltrative pulmonary disease, pericardial disease or myocardial infarction within 6 months prior to enrollment or left ventricular ejection fraction (LVEF) <40% within one month before randomization.
8. Ongoing or active systemic infection, active hepatitis A, B or C virus infection, or known human immunodeficiency virus (HIV) positivity.
9. Any other serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
10. Known allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib) or to any of the study medications, their analogues, or excipients in the various formulations of any agent.
11. Contraindication to dexamethasone or any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs, or intolerance to hydration due to pre-existing pulmonary or cardiac impairment.
12. Diagnosed or treated for another malignancy within 5 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
13. Patient has ≥ Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination within the 14 days prior to inclusion.
14. Participation in another interventional study within the 28 days before this study inclusion.
15. Patients refractory to carfilzomib or elotuzumab.
16. Primary plasma cell leukemia, systemic AL amyloidosis, Waldenström macroglobulinemia, rare Immunoglobulin M (IgM) multiple myeloma, POEMS syndrome, myelodysplasia
17. Allogeneic or autologous stem cell transplantation planned
18. Participants receiving any other investigational agents or received within 60 days
19. Pleural effusions requiring thoracocentesis within the 14 days prior the inclusion.
20. Ascites requiring puncture within the 14 days prior to inclusion.
21. Previous allogeneic transplantation
22. Uncontrolled hypertension or uncontrolled diabetes despite medication
23. Known hepatic cirrhosis
24. Severe autoimmune disease

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 3 years
  The proportion of patients having achieved at least partial response.

SECONDARY OUTCOMES:
Severe adverse events | 3 years
  Non-hematological grade 3 or more severe adverse events more or at least 70 percent

CONTACTS AND LOCATIONS:
Overall Officials: Raija Silvennoinen, MD, PhD, Principal Investigator — Helsinki University Central Hospital CCC Hematology
Locations (8):
- Finland (7):
  - Helsinki University Central Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Kymenlaakso Central Hospital, Kotka
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No